CLINICAL TRIAL: NCT00290680
Title: Phase I Trial of Bortezomib (VELCADE™) and Celecoxib in Patients With Advanced Solid Tumors
Brief Title: Bortezomib and Celecoxib in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000454922; MUSC-I065-341-03; MILLENNIUM-100825
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Bortezomib; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bortezomib
Drug: celecoxib

SUMMARY:
RATIONALE: Bortezomib and celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving bortezomib together with celecoxib may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib and celecoxib in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of bortezomib and celecoxib in patients with advanced solid tumors.

Secondary

* Determine the overall pattern of toxicities associated with this combination, including the emergence of any cumulative toxicities, during multiple courses of this regimen.
* Describe the response rate and duration of response or disease stability during therapy in the subset of patients with measurable disease.
* Assess changes in plasma/serum sphingosine-1-phosphate, ceramide, and other markers of the apoptotic pathway before and during therapy.

OUTLINE: This is a dose-escalation study.

Patients receive bortezomib IV on days 1, 4, 8, and 11 or days 1, 8, 15, 22, and 29 and oral celecoxib twice daily on days 1-21 or 1-42. Courses repeat every 21 or 42 days in the absence of disease progression or unacceptable toxicity. Patients are evaluated every 2 courses. Patients achieving complete response (CR) receive 2 additional courses of therapy beyond CR.

Cohorts of 3-6 patients receive escalating doses of bortezomib and celecoxib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologic or cytologic diagnosis of a malignant neoplasm (solid tumor) arising from any primary site with the exception of bone marrow or lymphoid tissue
* Recurrent or progressive disease after chemotherapy or radiotherapy

  * Chemotherapy or radiotherapy-naive disease allowed if patient is not a candidate for standard treatment either due to comorbidities or lack of willingness to undergo standard treatment
* Measurable disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 30 mL/min
* Bilirubin ≤ 2 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active concurrent invasive malignancy
* No peripheral neuropathy ≥ grade 2 within the past 14 days
* No hypersensitivity to bortezomib, boron, mannitol, any of the cyclooxygenase (COX-2) inhibitors, sulfa drugs, or other nonsteroidal anti-inflammatory drugs (NSAIDs)
* No active gastrointestinal (GI) ulcers OR history of GI bleeding resulting from prior therapy with NSAIDs

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since completion of prior radiotherapy
* No prior bortezomib
* No other concurrent investigational agents
* No concurrent chemotherapy, radiotherapy, or anticancer surgery
* No concurrent immune-enhancing therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose

SECONDARY OUTCOMES:
Response and disease progression by RECIST criteria before each course

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S. Kraft, MD, Study Chair — Medical University of South Carolina; Gustavo Leone, Study Chair — Medical University of South Carolina, Hollings Cancer Center
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Hayslip J, Chaudhary U, Green M, Meyer M, Dunder S, Sherman C, Salzer S, Kraft A, Montero AJ. Bortezomib in combination with celecoxib in patients with advanced solid tumors: a phase I trial. BMC Cancer. 2007 Dec 3;7:221. doi: 10.1186/1471-2407-7-221. PMID 18053191